CLINICAL TRIAL: NCT01299792
Title: Sonographic Measurement of Bladder Wall Thickness in Patients With Neurogenic Bladder Dysfunction Due to Spinal Cord Injury
Brief Title: Sonographic Measurement of Bladder Wall Thickness in Patients With Neurogenic Bladder Dysfunction
Status: Completed | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: 2009-07; EK900 (Registry Identifier: Ethic committee of Lucerne, Switzerland)
Record Dates: First submitted 2010-12-10; First posted 2011-02-18 (Estimated); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; urodynamics; ultrasound; neurogenic bladder dysfunction
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- one arm; neurogenic bladder dysfunction: evaluation of the clinical utility of bladder wall thickness as a diagnostic tool in patients with spinal cord injury
  Interventions: Other: sonographic measurement of bladder wall thickness

INTERVENTIONS:
Other: sonographic measurement of bladder wall thickness — measurement of bladder wall thickness by ultrasound at different filling states of the bladder during urodynamic investigation

SUMMARY:
Video-urodynamic investigations are regarded as the current standard diagnostics for neurogenic bladder dysfunction in patients with spinal cord injury. This examination is exact, but time consuming, costly and associated with the risk of urinary tract infection.

In patients with lower urinary tract symptoms due to benign prostate hyperplasia, sonographic measurement of bladder wall thickness has been demonstrated to be able to replace urodynamic testing for the diagnosis of infravesical obstruction.

Hypothesis: measurement of bladder wall thickness in patients with neurogenic bladder dysfunction due to spinal cord injury is closely related to the known risk factors for upper urinary tract deterioration (bladder compliance, detrusor leak point pressure) in this group of patients and can therefore replace urodynamic examination in selected cases.

ELIGIBILITY:
Inclusion Criteria:

* neurogenic bladder dysfunction due to spinal cord injury
* ability to understand German language
* willingness and capability to undergo urodynamic testing
* age > or = 18 years

Exclusion Criteria:

* acute urinary infection at the time of examination
* known bladder tumor or bladder stone
* age < 18 years
* not capable to understand aim and purpose of the examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: individuals with neurogenic bladder dysfunction due to spinal cord injury
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
correlation bladder wall thickness and detrusor compliance | calculated from maximum bladder filling
  measurement of detrusor compliance at maximum bladder volume; measurement of bladder wall thickness at maximum bladder volume

SECONDARY OUTCOMES:
correlation bladder wall thickness and maximum detrusor pressure | measurement at maximum bladder capacity
  correlation between bladder wall thickness and maximum detrusor pressure during the urodynamic storage phase

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Pannek, MD, Principal Investigator — Swiss Paraplegic Centre
Locations (1):
- Swiss paraplecic centre, Nottwil, Switzerland